CLINICAL TRIAL: NCT05290519
Title: Comparison of Plant-based or Animal-based Protein on Anthropocentric and Metabolic Parameters in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NTNU
Record Dates: First submitted 2022-03-01; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Abdominal; Glycation End Products, Advanced; Inflammation; Gut Microbiota
Keywords: advanced glycation end products; obesity; plant protein; inflammation; gut microbiota
MeSH Terms: conditions — Obesity, Abdominal; Inflammation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): plant protein for 4 weeks than animal protein for 4 weeks
  Interventions: Other: plant and animal protein
- Group B (Experimental): animal protein for 4 weeks than plant protein for 4 weeks
  Interventions: Other: plant and animal protein

INTERVENTIONS:
Other: plant and animal protein — plant protein: 2 bottle of black soy milk (400 mL/bottle) for 4 weeks animal protein: pork dished for 4 weeks

SUMMARY:
The investigators will try to evaluate the effects of substitution of dietary animal protein by black soybean milk (400 mL x 2) per day on anthropocentric and metabolic parameters in obese subjects.

DETAILED DESCRIPTION:
According to the survey by the Ministry of Health and Welfare, the proportion of obese male adolescents in Taiwan has been increasing year by year. Obesity is associated with chronic low-grade inflammation. Obese people prefer to intake foods containing higher levels of advanced glycation end products (AGEs). High intake of dietary AGEs (dAGEs) results in abdominal obesity, and shows positive correlation with body mass index (BMI) and waist circumference. When a large amount of AGEs accumulates in the body, inflammation usually occurs. Therefore, reducing dAGEs intake prevents the incidence of obesity, chronic diseases and aging. Black beans are high in protein. The black bean coats contain high level of anthocyanins. Previous studies demonstrated the biological functions of anthocyanins on blood lipid regulation, inflammation, and also inhibition of AGEs formation. Compared with meat (beef, pork, lamb, chicken, and seafood), the plant protein source, soy milk, under the same protein content showed significantly lower dAGE. In this study, the investigators will try to eveluate the effects of substitution of dietary animal protein by black soybean milk (400 mL x 2) per day on anthropocentric and metabolic parameters in obese subjects. This will be a randomized crossover interventional trial for 16 weeks: 0 to 4 weeks will be run-in period, 4 to 8 weeks and 12 to 16 weeks will be the soy milk or meat intervention period, and the between of two interventions (8 to 12 weeks) will be washout period. The body composition, blood pressure and AGE level will be measured. The blood, urine and feces sample will be collected for biochemical analysis and gut microbiome. The investigators expect the results could support the promotion of plant protein as part of dietary protein source to improve abnormal anthropometric and metabolic parameters in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 64 year male or female
* 27 <= BMI < 35 or waist circumference male >= 90 cm/female >= 80 cm
* fasting blood glucose: 100-125 mg/dL

Exclusion Criteria:

* Hypertension, cardiovascular disease, endocrine disease, acute and chronic liver and kidney disease, mental disease, binge or anorexia, or long-term drug use
* Consume probiotics, prebiotics, antibiotics or weight loss drugs regularly for the past month
* Try to lose weight and do resistance exercise regularly for the past month
* Allergic to soy products

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change from 4week blood advanced glycation end products level at 8 week | 4, 8 week
  blood AGEs level will be measured before and after intervention
change from 12 week blood advanced glycation end products level at 16 week | 12, 16 week
  blood AGEs level will be measured before and after intervention
change from 4 week blood leptin level at 8 week | 4, 8 week
  blood leptin level will be measured before and after intervention
change from 12 week blood leptin level at 16 week | 12, 16 week
  blood leptin level will be measured before and after intervention
change from 4 week blood adiponectin level at 8 week | 4, 8 week
  blood leptin level will be measured before and after intervention
change from 12 week blood adiponectin level at 16 week | 12, 16 week
  blood leptin level will be measured before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ju Yeh, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will be published in journals

REFERENCES:
- [Derived] Chang YH, Lee PN, Chen CH, Yang HY, Wu CH, Doong JY, Yeh WJ. Substituting animal protein with black soymilk reduces advanced glycation end product level and improves gut microbiota composition in obese prediabetic individuals: a randomized crossover intervention trial. Food Funct. 2025 Jan 2;16(1):195-206. doi: 10.1039/d4fo04717f. PMID 39651546